CLINICAL TRIAL: NCT03767517
Title: A Community Developed, Culturally-Based Palliative Care Tele-Consult Program for African American and White Rural Southern Elders With a Life Limiting Illness
Brief Title: A Culturally-Based Palliative Care Tele-consult Program for Rural Southern Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ronit Elk, Professor for the Division of Geriatrics, Gerontology, and Palliative Care; Associate Director for the Center for Palliative and Supportive Care, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB300002420; 1R01NR017181-01A1 (NIH); 5R01NR017181-05 (NIH)
Record Dates: First submitted 2018-10-29; First posted 2018-12-06 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Cardiac Disease; Pulmonary Disease; Neuro-Degenerative Disease; Renal Disease; Stroke; Sepsis; Hepatic Disease
MeSH Terms: conditions — Neoplasms; Heart Diseases; Lung Diseases; Kidney Diseases; Stroke; Sepsis; Digestive System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention (Experimental): Usual Care + Tele-consult Intervention
  Interventions: Other: Active Intervention
- Usual Care (Active Comparator): Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Active Intervention — Half of the patients will receive tele-consult program. Tele-consult intervention includes: initial consult and 2 follow up contacts. Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
  Arms: Active Intervention
Other: Usual Care — Half of the patients will receive usual care. Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
  Arms: Usual Care

SUMMARY:
Rural patients with life-limiting illness are at very high risk of not receiving appropriate care due to a lack of health professionals, long distances to treatment centers, and limited palliative care (PC) clinical expertise. Secondly, although culture strongly influences people's response to diagnosis, illness and treatment preferences, culturally-based care models are not currently available for most seriously-ill rural patients and their family caregivers. Lack of sensitivity to cultural differences may compromise PC for minority patients. The purpose of this study is to compare a culturally-based Tele-consult program to usual hospital care to determine whether a culturally-based PC Tele-consult program leads to lower symptom burden in hospitalized African American and White older adults with a life-limiting illness.

DETAILED DESCRIPTION:
The triple threat of rural geography, racial inequities, and older age hinders access to high quality PC for a significant proportion of Americans. Rural patients with life-limiting illness are at very high risk of not receiving appropriate care due to a lack of health professionals, long distances to treatment centers, and limited PC clinical expertise. Although culture strongly influences people's response to diagnosis, illness and treatment preferences, culturally-based care models are not currently available for most seriously-ill rural patients and their family caregivers. Lack of sensitivity to cultural differences may compromise PC for minority patients. The two major public health consequences of these problems are:

1. Access-Rural patients have sub-optimal or no access to PC. Despite significant nationwide growth, access to PC is grossly inadequate for the 60 million US citizens who live in rural or non-metropolitan areas. There is low PC use in rural and minority populations. As a result, rural patients experience significant suffering from uncontrolled symptoms that PC expertise could alleviate.
2. Acceptability-Even when palliative and hospice services are available, African Americans (AA), compared to Whites (W) are more likely to receive medically-ineffective, poor quality care due to a culturally-insensitive health care system and mistrust of health care providers. Making culturally competent PC available for diverse underserved and rural Americans is a national priority.

This community-developed, culturally based Teleconsult Intervention specifically targets the gaps of PC access and acceptability. It was developed by and for rural, Deep South AA and W patients and providers, and uses state-of-the-art telehealth methods, to provide PC consultation to hospitalized seriously-ill patients and family. Using National Consensus Project guidelines, and the culturally-based, community-developed PC Tele-consult intervention, a remote PC expert conducts a comprehensive PC patient assessment, in collaboration with local providers. Following interdisciplinary PC team review, the remote clinician communicates recommendations. Two additional structured follow up contacts at Day 3 and 6 ensure care coordination and smooth transitions that enable patients to receive guideline concurrent PC in their communities.

Aims of the study and Hypotheses:

Primary Aim: Determine whether a culturally-based PC Tele-consult program leads to lower symptom burden in hospitalized AA and W older adults with a life-limiting illness.

Hypothesis 1: Intervention patient participants receiving a culturally-based PC Tele-consult program will experience lower symptom burden on Day 7 post-consultation.

Secondary Aim: Determine whether a culturally-based PC Tele-consult program results in higher patient and caregiver quality of life, care satisfaction, and lower caregiver burden at Day 7 post-consultation, and lower resource use (hospital readmission, emergency visits) 30-days post-discharge.

Hypothesis 2: Intervention participants and their caregivers receiving a culturally-based PC Tele-consult program will experience higher patient and caregiver quality of life, care satisfaction, lower caregiver burden at Day 7 post consultation, and lower resource use (e.g. hospital admission, emergency visits) at 30 days after discharge.

Exploratory Aim: Explore mediators and moderators of patient symptom and caregiver burden outcomes.

ELIGIBILITY:
Inclusion Criteria:

* AA or W;
* 55 years old; has a condition which fits into one of 3 illness paradigms -cancer, chronic progressive, frailty.
* Clinician answers "no" to question: "Would you be surprised if this person died in the next 12 months?"
* Patient has a caregiver who has been involved in their care.
* Able to complete baseline interviews

Exclusion Criteria:

* Unable to complete baseline interviews;
* Currently receiving hospice care;
* No family member/caregiver.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Bakitas, DNSc, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - Russell Medical Center, Alexander City, Alabama
  - Anderson Regional Medical Center, Meridian, Mississippi
  - Highland Community Hospital, Picayune, Mississippi
  - Aiken Regional Medical Center, Aiken, South Carolina

REFERENCES:
- [Background] Watts KA, Gazaway S, Malone E, Elk R, Tucker R, McCammon S, Goldhagen M, Graham J, Tassin V, Hauser J, Rhoades S, Kagawa-Singer M, Wallace E, McElligott J, Kennedy R, Bakitas M. Community Tele-pal: A community-developed, culturally based palliative care tele-consult randomized controlled trial for African American and White Rural southern elders with a life-limiting illness. Trials. 2020 Jul 23;21(1):672. doi: 10.1186/s13063-020-04567-w. PMID 32703245
- [Background] Gazaway S, Bakitas M, Underwood F, Ekelem C, Duffie M, McCormick S, Heard V, Colvin A, Elk R. Community Informed Recruitment: A Promising Method to Enhance Clinical Trial Participation. J Pain Symptom Manage. 2023 Jun;65(6):e757-e764. doi: 10.1016/j.jpainsymman.2023.02.319. Epub 2023 Mar 5. PMID 36871774
- [Background] Allen Watts K, Malone E, Dionne-Odom JN, McCammon S, Currie E, Hicks J, Tucker RO, Wallace E, Elk R, Bakitas M. Can you hear me now?: Improving palliative care access through telehealth. Res Nurs Health. 2021 Feb;44(1):226-237. doi: 10.1002/nur.22105. Epub 2021 Jan 4. PMID 33393704
- [Background] Gazaway S, Bakitas MA, Elk R, Eneanya ND, Dionne-Odom JN. Engaging African American family Caregivers in Developing a Culturally-responsive Interview Guide: A Multiphase Process and Approach. J Pain Symptom Manage. 2022 Jun;63(6):e705-e711. doi: 10.1016/j.jpainsymman.2022.02.331. Epub 2022 Mar 3. PMID 35247583
- [Background] Gazaway S, Odom JN, Herbey I, Armstrong M, Underwood F, Heard TV, Allen A, Ekelem C, Bakitas MA, Elk R. Cultural Values Influence on Rural Family Caregivers' Decision-Making for Ill Older Adult Loved Ones. J Pain Symptom Manage. 2024 Jul;68(1):86-95. doi: 10.1016/j.jpainsymman.2024.04.012. Epub 2024 Apr 18. PMID 38641135
- [Result] Gazaway, S., Bakitas, MA., Underwood, F., Ekelem, C., Duffie, M., McCormick, S., Heard, V., Massey,. L., Allen, A., Tucker, R., McCammon, S., Goldhagen, M., Hauser, J., McElwain, L., Kennedy, R., Azuero, A., & Elk, R. Community Tele-Pal RCT Videoconsultation for Rural White and Black Inpatients: Caregiver Outcomes. American Association of Hospice and Palliative Medicine and the Hospice and Palliative Nurses Association Annual Assembly 2024.
- [Result] Bakitas, MA., Gazaway, S., Underwood, F., Ekelem, C., Duffie, M., McCormick, S., Heard, V., Massey,. L., Allen, A., Tucker, R., McCammon, S., Goldhagen, M., Hauser, J., McElwain, L., Kennedy, R., Azuero, A., & Elk, R. Community Tele-Pal RCT Videoconsultation for Rural White and Black Inpatients: Patient Outcomes. American Association of Hospice and Palliative Medicine and the Hospice and Palliative Nurses Association Annual Assembly 2024.
- [Derived] Bakitas MA, Gazaway S, Underwood F, Ekelem C, Heard VT, Kennedy R, Azuero A, Tucker R, McCammon S, Hauser JM, McElwain L, Elk R. Palliative Video Consultation and Symptom Distress Among Rural Inpatients: A Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2519426. doi: 10.1001/jamanetworkopen.2025.19426. PMID 40632537

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patient and Caregivers were considered enrolled. The patients were not enrolled without an active caregiver. They were only given one study Identification number.
Period: Overall Study
Arm/Group | Active Intervention | Usual Care
Started | 105 | 104
Patient/Caregiver Breakdown | 105 (105 Active Intervention patient participants and 105 caregiver participants were enrolled in this study.) | 104 (104 Usual Care Patient participants and 104 Caregiver participants were enrolled in the study.)
Completed | 87 (There were 36 patient/caregiver did not complete the study in the active intervention group.) | 91 (There were 26 patient/caregiver that did not complete the usual care study.)
Not Completed | 18 | 13
Not completed — Lost to Follow-up | 16 | 10
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Population: There are 105 patient participants and 105 caregiver participants in the active intervention and the participants were analyzed in their respective groups. There are 104 patient participants and 104 caregiver participants and the participants were analyzed in their respective groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention | Usual Care | Total
Number analyzed (Participants) | 210 | 208 | 418
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There are 105 patient participants and 105 caregiver participants in the active intervention and the participants were analyzed in their respective groups. There are 104 patient participants and 104 caregiver participants and the participants were analyzed in their respective groups.
  years
    Patients: number analyzed (Participants) | 105 | 104 | 209
    Patients | 72.9 (8.7) | 73.7 (7.7) | 73.3 (8.2)
    Caregivers: number analyzed (Participants) | 105 | 104 | 209
    Caregivers | 61.5 (14.6) | 58.6 (15.5) | 60.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: # of caregivers in USUAL CARE were lost to f/u
  Participants
    Patients: number analyzed (Participants) | 105 | 104 | 209
    Patients: Female | 53 | 67 | 120
    Patients: Male | 52 | 37 | 89
    Caregivers: number analyzed (Participants) | 105 | 101 | 206
    Caregivers: Female | 83 | 72 | 155
    Caregivers: Male | 22 | 29 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The ethnicity measure was assessed only for patients enrolled in the study. Population: There are 105 patient participants in the active intervention and There are 104 patient participants in usual care.
  Participants
    Patient: number analyzed (Participants) | 105 | 104 | 209
    Patient: Hispanic or Latino | 0 | 0 | 0
    Patient: Not Hispanic or Latino | 105 | 104 | 209
    Patient: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: There are 105 patient participants and 105 caregiver participants in the active intervention and the participants were analyzed in their respective groups. There are 104 patient participants and 104 caregiver participants and the participants were analyzed in their respective groups.
  Participants
    Patients: number analyzed (Participants) | 105 | 104 | 209
    Patients: American Indian or Alaska Native | 0 | 0 | 0
    Patients: Asian | 0 | 0 | 0
    Patients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patients: Black or African American | 30.0 | 28.0 | 58
    Patients: White | 75.0 | 76.0 | 151
    Patients: More than one race | 0 | 0 | 0
    Patients: Unknown or Not Reported | 0 | 0 | 0
    Caregivers: number analyzed (Participants) | 105 | 104 | 209
    Caregivers: American Indian or Alaska Native | 0 | 0 | 0
    Caregivers: Asian | 0 | 0 | 0
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregivers: Black or African American | 29.0 | 27.0 | 56
    Caregivers: White | 76.0 | 73.0 | 149
    Caregivers: More than one race | 0 | 0 | 0
    Caregivers: Unknown or Not Reported | 0 | 4.0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 210 | 208 | 418

OUTCOME MEASURES:

1. Primary Outcome: Patient Symptom Burden (Edmonton Symptom Assessment Scale [ESAS])
Description: Change from baseline in patient-reported symptom burden measured using the Edmonton Symptom Assessment Scale (ESAS) at baseline; change from baseline measured using the ESAS at 7 days post-baseline. Each item is scored using: 0-10 (0= no pain; 10= worst possible pain), yielding a total score between 0 and 90. A higher value represents the worse possible outcome. Higher score indicates higher symptom burden.
Time Frame: baseline and 7 days post-baseline and 30 days post-baseline
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
score on a scale
  baseline | 35.1 (0.9) | 34.6 (0.9)
  Day 7 | 38.6 (0.9) | 38 (0.9)
  Day 30 | 40.5 (0.9) | 39.4 (0.9)

2. Secondary Outcome: The Mean Percentage of Caregivers Who Responded Very Satisfied/Satisfied to the Family Satisfaction With Care (FAMCARE-2) Survey.
Description: Change from baseline measured using FAMCARE-2 at 7 days post-baseline. Each item was scored on a Likert scale of VS (very satisfied), S (satisfied), U (undecided), D (dissatisfied), VD (very dissatisfied), or NA (not applicable), which was then dichotomized into very satisfied/satisfied and undecided/dissatisfied/very dissatisfied. The mean percentages in these dichotomized categories was calculated along with the standard error of the mean. A repeated measures generalized linear mixed model was used to calculate the estimated marginal means (least squares means) and associated standard errors at each time point for the intervention and usual care groups. The higher mean percentage of the population that responded very satisfied/ satisfied equals a better outcome.
Time Frame: baseline and 7 days post-baseline and 30 days post baseline
Population: The participants number analyzed in one or more rows differ from the overall number analyzed due to participants choosing not to answer certain questions from baseline to day 30.
Measure: Number; unit: percentage of participants
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
percentage of participants
  Baseline Patient Comfort-Very satisfied/ Satisfied: number analyzed (Participants) | 101 | 98
  Baseline Patient Comfort-Very satisfied/ Satisfied | 76.2 | 78.6
  Baseline Patient Comfort Undecided/dissatisfied/very dissatisfied: number analyzed (Participants) | 101 | 98
  Baseline Patient Comfort Undecided/dissatisfied/very dissatisfied | 23.8 | 21.4
  Day 7 Patient Comfort-Very satisfied/ Satisfied: number analyzed (Participants) | 91 | 92
  Day 7 Patient Comfort-Very satisfied/ Satisfied | 85.7 | 84.8
  Day 7 Patient Comfort-Undecided/Dissatisfied/very dissatisfied: number analyzed (Participants) | 91 | 92
  Day 7 Patient Comfort-Undecided/Dissatisfied/very dissatisfied | 14.3 | 15.2
  Day 30 Patient Comfort Very satisfied/Satisfied: number analyzed (Participants) | 87 | 90
  Day 30 Patient Comfort Very satisfied/Satisfied | 94.3 | 90
  Day 30 Patient Comfort Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 87 | 90
  Day 30 Patient Comfort Undecided/Dissatisfied/Very Dissatisfied | 5.7 | 10
  Baseline-Conditions and progress explained-Very Satisfied/Satisfied: number analyzed (Participants) | 98 | 91
  Baseline-Conditions and progress explained-Very Satisfied/Satisfied | 70.8 | 71.9
  Baseline Condition and Progress explained-Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 98 | 91
  Baseline Condition and Progress explained-Undecided/Dissatisfied/Very Dissatisfied | 29.2 | 28.1
  Day 7 Conditions and Progress explained-Very Satisfied/Satisfied: number analyzed (Participants) | 88 | 89
  Day 7 Conditions and Progress explained-Very Satisfied/Satisfied | 80.6 | 85.4
  Day 7 Conditions and Progress explained- Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 88 | 89
  Day 7 Conditions and Progress explained- Undecided/Dissatisfied/Very Dissatisfied | 19.4 | 14.6
  Day 30-Conditions and Progress Explained- Very Satisfied/Satisfied: number analyzed (Participants) | 85 | 89
  Day 30-Conditions and Progress Explained- Very Satisfied/Satisfied | 90.6 | 92.7
  Day 30 Conditions and Progress Explained-Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 85 | 89
  Day 30 Conditions and Progress Explained-Undecided/Dissatisfied/Very Dissatisfied | 9.4 | 7.3
  Baseline-Information on Side Effects Very Satisfied/Satisfied: number analyzed (Participants) | 99 | 93
  Baseline-Information on Side Effects Very Satisfied/Satisfied | 77 | 72.8
  Baseline-Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 99 | 93
  Baseline-Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied | 23 | 27.2
  Day 7 Information on Side Effects Very Satisfied/Satisfied: number analyzed (Participants) | 86 | 88
  Day 7 Information on Side Effects Very Satisfied/Satisfied | 87.2 | 78.5
  Day 7 Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 86 | 88
  Day 7 Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied | 12.8 | 21.5
  Day 30 Information on Side Effects/Very Satisfied/Satisfied: number analyzed (Participants) | 85 | 88
  Day 30 Information on Side Effects/Very Satisfied/Satisfied | 91.3 | 86.4
  Day 30 Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 85 | 88
  Day 30 Information on Side Effects/ Undecided/Dissatisfied/Very Dissatisfied | 8.7 | 13.6
  Baseline-Respect for Dignity/ Very Satisfied/Satisfied: number analyzed (Participants) | 101 | 95
  Baseline-Respect for Dignity/ Very Satisfied/Satisfied | 88.1 | 87.4
  Baseline-Respect for Dignity/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 101 | 95
  Baseline-Respect for Dignity/ Undecided/Dissatisfied/Very Dissatisfied | 11.9 | 12.6
  Day 7-Respect for Dignity/ Very Satisfied/Satisfied: number analyzed (Participants) | 89 | 89
  Day 7-Respect for Dignity/ Very Satisfied/Satisfied | 84.3 | 88.8
  Day 7-Respect for Dignity/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 89 | 89
  Day 7-Respect for Dignity/Undecided/Dissatisfied/Very Dissatisfied | 15.7 | 11.2
  Day 30 Respect for Dignity/Very Satisfied/Satisfied: number analyzed (Participants) | 86 | 89
  Day 30 Respect for Dignity/Very Satisfied/Satisfied | 91.9 | 93.3
  Day 30 Respect for Dignity/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 86 | 89
  Day 30 Respect for Dignity/ Undecided/Dissatisfied/Very Dissatisfied | 8.1 | 6.7
  Baseline Meetings with Care Team/ Very Satisfied/ Satisfied: number analyzed (Participants) | 89 | 87
  Baseline Meetings with Care Team/ Very Satisfied/ Satisfied | 64.4 | 68.2
  Baseline Meetings with Care Team/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 89 | 87
  Baseline Meetings with Care Team/ Undecided/Dissatisfied/Very Dissatisfied | 35.6 | 31.8
  Day 7 Meetings with Care Team/Very Satisfied/Satisfied: number analyzed (Participants) | 83 | 84
  Day 7 Meetings with Care Team/Very Satisfied/Satisfied | 85.7 | 83
  Day 7 Meeting with Care Team/ Undecided/Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 83 | 84
  Day 7 Meeting with Care Team/ Undecided/Dissatisfied/ Very Dissatisfied | 14.3 | 17
  Day 30-Meetings with Care Team/Satisfied/Very Satisfied: number analyzed (Participants) | 81 | 85
  Day 30-Meetings with Care Team/Satisfied/Very Satisfied | 87.2 | 89.7
  Day 30 Meetings with Care Team/Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 81 | 85
  Day 30 Meetings with Care Team/Undecided/ Dissatisfied/Very Dissatisfied | 12.8 | 10.3
  Baseline Speed of Treatment/Very Satisfied/Satisfied: number analyzed (Participants) | 102 | 98
  Baseline Speed of Treatment/Very Satisfied/Satisfied | 71 | 62.4
  Baseline Speed of Treatment/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 102 | 98
  Baseline Speed of Treatment/ Undecided/ Dissatisfied/Very Dissatisfied | 29 | 37.6
  Day 7 Speed of Treatment/ Very Satisfied/Satisfied: number analyzed (Participants) | 90 | 89
  Day 7 Speed of Treatment/ Very Satisfied/Satisfied | 78.8 | 81.7
  Day 7 Speed of Treatment/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 90 | 89
  Day 7 Speed of Treatment/ Undecided/ Dissatisfied/ Very Dissatisfied | 21.2 | 18.3
  Day 30 Speed of Treatment/ Very Satisfied/Satisfied: number analyzed (Participants) | 87 | 89
  Day 30 Speed of Treatment/ Very Satisfied/Satisfied | 91.6 | 87.1
  Day 30 Speed of Treatment/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 87 | 89
  Day 30 Speed of Treatment/ Undecided/ Dissatisfied/ Very Dissatisfied | 8.4 | 12.9
  Baseline Attention to Symptom description/ Very satisfied/Satisfied: number analyzed (Participants) | 102 | 96
  Baseline Attention to Symptom description/ Very satisfied/Satisfied | 80.6 | 74.8
  Baseline Attentions to Symptom description/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 102 | 96
  Baseline Attentions to Symptom description/ Undecided/ Dissatisfied/Very Dissatisfied | 19.4 | 25.2
  Day 7 Attention to Symptom description/ Very Satisfied/ Satisfied: number analyzed (Participants) | 91 | 89
  Day 7 Attention to Symptom description/ Very Satisfied/ Satisfied | 82.4 | 84.1
  Day 7 Attention to Symptom Description/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 91 | 89
  Day 7 Attention to Symptom Description/ Undecided/ Dissatisfied/ Very Dissatisfied | 17.6 | 15.9
  Day 30 Attention to Symptom Description/ Very Satisfied/ Satisfied: number analyzed (Participants) | 86 | 88
  Day 30 Attention to Symptom Description/ Very Satisfied/ Satisfied | 92.8 | 94.1
  Day 30 Attention to Symptom Description/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 86 | 88
  Day 30 Attention to Symptom Description/ Undecided/ Dissatisfied/ Very Dissatisfied | 7.2 | 5.9
  Baseline Physical Needs Met/ Very Satisfied/ Satisfied: number analyzed (Participants) | 101 | 97
  Baseline Physical Needs Met/ Very Satisfied/ Satisfied | 84.8 | 83.1
  Baseline Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 101 | 97
  Baseline Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied | 15.2 | 16.9
  Day 7 Physical Needs Met/ Very Satisfied/ Satisfied: number analyzed (Participants) | 89 | 91
  Day 7 Physical Needs Met/ Very Satisfied/ Satisfied | 85.1 | 85.3
  Day 7 Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 89 | 91
  Day 7 Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied | 14.9 | 14.7
  Day 30 Physical Needs Met/ Very Satisfied/ Satisfied: number analyzed (Participants) | 87 | 89
  Day 30 Physical Needs Met/ Very Satisfied/ Satisfied | 92.8 | 93.4
  Day 30 Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 87 | 89
  Day 30 Physical Needs Met/ Undecided/ Dissatisfied/ Very Dissatisfied | 7.2 | 6.6
  Baseline Availability of Care Team/ Very Satisfied/ Satisfied: number analyzed (Participants) | 100 | 95
  Baseline Availability of Care Team/ Very Satisfied/ Satisfied | 75.5 | 73.9
  Baseline Availability of Care Team Undecided/Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 100 | 95
  Baseline Availability of Care Team Undecided/Dissatisfied/ Very Dissatisfied | 24.5 | 26.1
  Day 7 Availability of Care Team/Very Satisfied/ Satisfied: number analyzed (Participants) | 87 | 89
  Day 7 Availability of Care Team/Very Satisfied/ Satisfied | 85.4 | 87.7
  Day 7 Availability of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 87 | 89
  Day 7 Availability of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied | 14.6 | 12.3
  Day 30 Availability of Care Team/ Very Satisfied/ Satisfied: number analyzed (Participants) | 84 | 88
  Day 30 Availability of Care Team/ Very Satisfied/ Satisfied | 90.8 | 94.5
  Day 30 Availability of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 84 | 88
  Day 30 Availability of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied | 9.2 | 5.5
  Baseline Emotional Support to Family/Very Satisfied/Satisfied: number analyzed (Participants) | 89 | 87
  Baseline Emotional Support to Family/Very Satisfied/Satisfied | 76 | 79.4
  Baseline Emotional Support to Family Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 89 | 87
  Baseline Emotional Support to Family Undecided/ Dissatisfied/ Very Dissatisfied | 24 | 20.6
  Day 7 Emotional Support of Family/Very Satisfied/ Satisfied: number analyzed (Participants) | 85 | 86
  Day 7 Emotional Support of Family/Very Satisfied/ Satisfied | 81.2 | 85
  Day 7 Emotional Support to Family/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 85 | 86
  Day 7 Emotional Support to Family/ Undecided/ Dissatisfied/ Very Dissatisfied | 18.8 | 15
  Day 30 Emotional Support to Family/ Very Satisfied/ Satisfied: number analyzed (Participants) | 85 | 86
  Day 30 Emotional Support to Family/ Very Satisfied/ Satisfied | 90.9 | 91.3
  Day 30 Emotional Support to Family Undecided/Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 85 | 86
  Day 30 Emotional Support to Family Undecided/Dissatisfied/ Very Dissatisfied | 9.1 | 8.7
  Baseline Practical Assistance/Very Satisfied/ Satisfied: number analyzed (Participants) | 65 | 76
  Baseline Practical Assistance/Very Satisfied/ Satisfied | 86.2 | 78.9
  Baseline Practical Assistance/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 65 | 76
  Baseline Practical Assistance/ Undecided/ Dissatisfied/ Very Dissatisfied | 13.8 | 21.1
  Day 7 Practical Assistance/Very Satisfied/ Satisdfied: number analyzed (Participants) | 65 | 67
  Day 7 Practical Assistance/Very Satisfied/ Satisdfied | 80 | 85.1
  Day 7 Practical Assistance/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 65 | 67
  Day 7 Practical Assistance/Undecided/Dissatisfied/Very Dissatisfied | 20 | 14.9
  Day 30 Practical Assistance Very Satisfied/ Satisfied: number analyzed (Participants) | 58 | 68
  Day 30 Practical Assistance Very Satisfied/ Satisfied | 84.5 | 85.3
  Day 30 Practical Assistance Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 58 | 68
  Day 30 Practical Assistance Undecided/ Dissatisfied/Very Dissatisfied | 15.5 | 14.7
  Baseline Doctors Attention to Symptoms/Very Satisfied/Satisfied: number analyzed (Participants) | 101 | 93
  Baseline Doctors Attention to Symptoms/Very Satisfied/Satisfied | 80.2 | 80.6
  Baseline Doctors Attention to Symptoms/ Undecided/Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 101 | 93
  Baseline Doctors Attention to Symptoms/ Undecided/Dissatisfied/ Very Dissatisfied | 19.8 | 19.4
  Day 7 Doctors Attention to Symptoms/ Very Satisfied/Satisfied: number analyzed (Participants) | 89 | 87
  Day 7 Doctors Attention to Symptoms/ Very Satisfied/Satisfied | 84.3 | 85.1
  Day 7 Doctors Attention to Symptoms/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 89 | 87
  Day 7 Doctors Attention to Symptoms/ Undecided/Dissatisfied/Very Dissatisfied | 15.7 | 14.9
  Day 30 Doctors Attention to Symptoms/Very Satisfied/Satisfied: number analyzed (Participants) | 84 | 87
  Day 30 Doctors Attention to Symptoms/Very Satisfied/Satisfied | 92.9 | 88.5
  Day 30 Doctors Attention to Symptoms/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 84 | 87
  Day 30 Doctors Attention to Symptoms/Undecided/Dissatisfied/Very Dissatisfied | 7.1 | 11.5
  Baseline Family Included/Very Satisfied/Satisfied: number analyzed (Participants) | 101 | 90
  Baseline Family Included/Very Satisfied/Satisfied | 81.2 | 75.6
  Baseline Family Included/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 101 | 90
  Baseline Family Included/ Undecided/Dissatisfied/Very Dissatisfied | 18.8 | 24.4
  Day 7 Family Included/ Very Satisfied/Satisfied: number analyzed (Participants) | 89 | 89
  Day 7 Family Included/ Very Satisfied/Satisfied | 85.4 | 86.5
  Day 7 Family Included/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 89 | 89
  Day 7 Family Included/ Undecided/Dissatisfied/Very Dissatisfied | 14.6 | 13.5
  Day 30 Family Included/ Very Satisfied/Satisfied: number analyzed (Participants) | 83 | 88
  Day 30 Family Included/ Very Satisfied/Satisfied | 89.2 | 92
  Day 30 Family Included/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 83 | 88
  Day 30 Family Included/ Undecided/ Dissatisfied/ Very Dissatisfied | 10.8 | 8
  Baseline Info about managing symptoms/ Very Satisfied/ Satisfied: number analyzed (Participants) | 79 | 74
  Baseline Info about managing symptoms/ Very Satisfied/ Satisfied | 68.6 | 69.6
  Baseline Info about managing symptoms/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 79 | 74
  Baseline Info about managing symptoms/ Undecided/ Dissatisfied/Very Dissatisfied | 31.4 | 30.4
  Day 7 Info about managing symptoms/Very Satisfied/Satisfied: number analyzed (Participants) | 68 | 70
  Day 7 Info about managing symptoms/Very Satisfied/Satisfied | 83.8 | 81.2
  Day 7 Info about managing symptoms/ Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 68 | 70
  Day 7 Info about managing symptoms/ Undecided/Dissatisfied/Very Dissatisfied | 16.2 | 18.8
  Day 30 Info about managing symptoms/ Very Satisfied/Satisfied: number analyzed (Participants) | 63 | 80
  Day 30 Info about managing symptoms/ Very Satisfied/Satisfied | 84.9 | 92
  Day 30 Info about managing symptoms/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 63 | 80
  Day 30 Info about managing symptoms/ Undecided/ Dissatisfied/Very Dissatisfied | 15.1 | 8
  Baseline Effectiveness of Care Team/ Very Satisfied/Satisfied: number analyzed (Participants) | 100 | 95
  Baseline Effectiveness of Care Team/ Very Satisfied/Satisfied | 81.4 | 78.9
  Baseline Effectiveness of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 100 | 95
  Baseline Effectiveness of Care Team/ Undecided/ Dissatisfied/ Very Dissatisfied | 18.6 | 21.1
  Day 7 Effectiveness of Care Team/Very Satisfied/Satisfied: number analyzed (Participants) | 90 | 89
  Day 7 Effectiveness of Care Team/Very Satisfied/Satisfied | 83.6 | 90.7
  Day 7 Effectiveness of Care Team/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 90 | 89
  Day 7 Effectiveness of Care Team/ Undecided/ Dissatisfied/Very Dissatisfied | 16.4 | 9.3
  Day 30 Effectiveness of Care Team/Very Satisfied/Satisfied: number analyzed (Participants) | 85 | 89
  Day 30 Effectiveness of Care Team/Very Satisfied/Satisfied | 91.7 | 92.4
  Day 30 Effectiveness of Care Team/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 85 | 89
  Day 30 Effectiveness of Care Team/Undecided/Dissatisfied/Very Dissatisfied | 8.3 | 7.6
  Baseline Response to Changes/Very Satisfied/Satisfied: number analyzed (Participants) | 100 | 94
  Baseline Response to Changes/Very Satisfied/Satisfied | 77 | 77.7
  Baseline Response to Changes/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 100 | 94
  Baseline Response to Changes/Undecided/Dissatisfied/Very Dissatisfied | 23 | 22.3
  Day 7 Response to Changes/Very Satisfied/ Satisfied: number analyzed (Participants) | 87 | 86
  Day 7 Response to Changes/Very Satisfied/ Satisfied | 83.9 | 89.5
  Day 7 Response to Changes/ Undecided/ Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 87 | 86
  Day 7 Response to Changes/ Undecided/ Dissatisfied/Very Dissatisfied | 16.1 | 10.5
  Day 30 Response to Changes/Very Satisfied/ Satisfied: number analyzed (Participants) | 83 | 88
  Day 30 Response to Changes/Very Satisfied/ Satisfied | 92.8 | 92
  Day 30 Response to Changes/ Undecided/Dissatisfied/ Very Dissatisfied: number analyzed (Participants) | 83 | 88
  Day 30 Response to Changes/ Undecided/Dissatisfied/ Very Dissatisfied | 7.2 | 8
  Baseline Emotional Support to Patient/Very Satisfied/Satisfied: number analyzed (Participants) | 99 | 90
  Baseline Emotional Support to Patient/Very Satisfied/Satisfied | 79.8 | 80
  Baseline Emotional Support to Patient/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 99 | 90
  Baseline Emotional Support to Patient/Undecided/Dissatisfied/Very Dissatisfied | 20.2 | 20
  Day 7 Emotional Support to Patient/Very Satisfied/Satisfied: number analyzed (Participants) | 87 | 88
  Day 7 Emotional Support to Patient/Very Satisfied/Satisfied | 89.7 | 87.5
  Day 7 Emotional Support to Patient/Undecided/Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 87 | 88
  Day 7 Emotional Support to Patient/Undecided/Dissatisfied/Very Dissatisfied | 10.3 | 12.5
  Day 30 Emotional Support to Patient/Very Satisfied/Satisfied: number analyzed (Participants) | 83 | 88
  Day 30 Emotional Support to Patient/Very Satisfied/Satisfied | 89.2 | 90.9
  Day 30 Emotional Support to Patient/Undecided Dissatisfied/Very Dissatisfied: number analyzed (Participants) | 83 | 88
  Day 30 Emotional Support to Patient/Undecided Dissatisfied/Very Dissatisfied | 10.8 | 9.1

3. Secondary Outcome: Patient Quality of Life (Patient-Reported Outcomes Measurement Information System Global Health-10 [PROMIS Global Health-10])
Description: Change from baseline in patient-reported quality of life using the Patient-Reported Outcomes Measurement Information System Global Health-10 (PROMIS Global Health-10) at baseline; change from baseline measured using the PROMIS Health-10 at 7 days post-baseline. Items 1-6 are scored using: 1-5 (1=poor; 5=excellent). Item 7 is scored using 1-5 (1= not at all; 5= completely). Item 8 is scored using 1-5 (1= always; 5=never). Item 9 is scored using 1-5 (1=very severe; 5=none). Item 10 is scored using 0-10 (0=no pain; 10=worst pain imaginable).Items were summed , then scaled to T-scores (which would have a mean of 50 and standard deviation of 10 in the general adult population) using published procedures from Health Measures, with higher scores representing better health. As the PROMIS Global Health is scaled relative to the referent general population, there are no minimum and maximum values published.
Time Frame: baseline and 7 days post-baseline
Population: The number of patients changed because of not completing the study.
Measure: Mean (Standard Error); unit: scaled to T-Scores
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
scaled to T-Scores
  Baseline Physical Health | 35.1 (0.9) | 34.6 (0.9)
  Day 7 Physical Health: number analyzed (Participants) | 94 | 95
  Day 7 Physical Health | 38.6 (0.9) | 38 (0.9)
  Baseline Mental Health: number analyzed (Participants) | 104 | 104
  Baseline Mental Health | 45.5 (0.8) | 43.7 (0.8)
  Day 7 Mental Health: number analyzed (Participants) | 95 | 95
  Day 7 Mental Health | 45.7 (0.8) | 44 (0.8)

4. Secondary Outcome: Caregiver Quality of Life (Patient-Reported Outcomes Measurement Information System Global Health-10 [PROMIS Global Health-10])
Description: Change from baseline in caregiver-reported quality of life using the Patient-Reported Outcomes Measurement Information System Global Health-10 (PROMIS Global Health-10) at baseline; change from baseline measured using the PROMIS Global Health-10 at 7 days post-baseline. Items 1-6 are scored using: 1-5 (1=poor; 5=excellent). Item 7 is scored using 1-5 (1= not at all; 5= completely). Item 8 is scored using 1-5 (1= always; 5=never). Item 9 is scored using 1-5 (1=very severe; 5=none). Item 10 is scored using 0-10 (0=no pain; 10=worst pain imaginable).Items were summed , then scaled to T-scores (which would have a mean of 50 and standard deviation of 10 in the general adult population) using published procedures from Health Measures, with higher scores representing better health. As the PROMIS Global Health is scaled relative to the referent general population, there are no minimum and maximum values published.
Time Frame: Baseline and 7 days post-Baseline
Population: The number of Caregivers changed at Day 7.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 104 | 101
score on a scale
  Baseline Physical Health | 48.5 (0.9) | 47.6 (0.9)
  Day 7 Physical Health: number analyzed (Participants) | 94 | 95
  Day 7 Physical Health | 50.9 (0.9) | 49.4 (0.9)
  Baseline Mental Health: number analyzed (Participants) | 102 | 101
  Baseline Mental Health | 50 (0.7) | 47.7 (0.7)
  Day 7 Mental Health: number analyzed (Participants) | 94 | 95
  Day 7 Mental Health | 49.6 (0.7) | 48.3 (0.7)

5. Secondary Outcome: Caregiver Burden Scale (Montgomery Borgatta Caregiver Burden Scale [MBCB])
Description: Change from baseline in caregiver-reported burden using the Montgomery Borgatta Caregiver Burden Scale (MBCB) at baseline; change from baseline measured using the MBCB at 7 days post-baseline. This scale contains a total of 14 questions and 5 Likert scale responses (a lot less, a little less, the same, a little more, or a lot more). Caregiver burden will be quantified by three subscales; objective, subjective and demand burdens. Objective burden is measured by 6 questions (total score between 0-30), subjective burden is measured by 4 questions (total score between 4-20), and demand burden is measured by 4 questions (total score between 4-20).
Time Frame: Baseline and 7 days post-Baseline
Population: The number analyzed in one or more rows differ from the overall number analyzed because some of the participants failed to answer questions during data collection.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
score on a scale
  Baseline Objective Burden: number analyzed (Participants) | 103 | 97
  Baseline Objective Burden | 19.5 (0.3) | 19.9 (0.3)
  Day 7 Objective Burden: number analyzed (Participants) | 88 | 93
  Day 7 Objective Burden | 19.1 (0.3) | 19.4 (0.3)
  Baseline Subjective Burden: number analyzed (Participants) | 103 | 98
  Baseline Subjective Burden | 13.4 (0.3) | 13.1 (0.3)
  Day 7 Subjective Burden: number analyzed (Participants) | 78 | 85
  Day 7 Subjective Burden | 11.9 (0.3) | 11.6 (0.3)
  Baseline Demand Burden: number analyzed (Participants) | 96 | 88
  Baseline Demand Burden | 12.1 (0.3) | 11.8 (0.3)
  Day 7 Demand Burden: number analyzed (Participants) | 72 | 78
  Day 7 Demand Burden | 11 (0.3) | 10.8 (0.3)

6. Secondary Outcome: Resource Use
Description: Patient resource use (e.g., number of hospital readmissions, and number of Emergency Department [ED] visits) within 30 days after enrollment.
Time Frame: 30 days post-Baseline
Population: Some participants reported that they were not sure which was considered missing data for analysis.
Measure: Mean (Standard Error); unit: count the number of visits
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 90 | 91
count the number of visits
  Number of ER visits | 0.19 (0.06) | 0.16 (0.05)
  Number of Hospital Re-admissions | 0.2 (0.06) | 0.14 (0.04)

7. Secondary Outcome: The Mean Percentage of Caregivers Who Responded Completely/Quite a Bit to the Patient Satisfaction With Care (Feeling Heard and Understood) Survey.
Description: Change from baseline in patient-reported satisfaction with care using the Feeling Heard and Understood questionnaire at baseline; change from baseline using the Feeling Heard and Understood questionnaire at 7 days post-baseline. Likert scale using: completely, quite a bit, moderately, slightly, not at all. Which was then dichotomized into completely/quite-a-bit and moderately/slightly/not at all. The mean percentage of participants in these dichotomized categories were calculated along with the standard error of the mean. The higher mean percentage of the population that responded completely/ quite a bit equals a better outcome.
Time Frame: Baseline and 7 days post-Baseline
Population: Nine of the participants dropped out of the study by Day 7.
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 104 | 104
percentage of participants
  Baseline Completely/Quite a bit | 76.9 (4.1) | 76.9 (4.1)
  Day 7 Completely/ Quite a Bit | 88.4 (3.3) | 90.5 (3)
  Baseline Moderately/Slightly/Not at all: number analyzed (Participants) | 95 | 95
  Baseline Moderately/Slightly/Not at all | 23.1 (4.1) | 23.1 (4.1)
  Day 7 Moderately/Slightly/Not at all: number analyzed (Participants) | 95 | 95
  Day 7 Moderately/Slightly/Not at all | 11.6 (3.3) | 9.5 (3)

8. Other Pre Specified Outcome: Exploratory Aim 1a. Patient Symptom Burden (Edmonton Symptom Assessment Scale [ESAS])
Description: Patient symptom burden measured by Edmonton Symptom Assessment Scale [ESAS] mediated and/or moderated by hospitalist/clinician implementation of palliative care recommendations. Implementation of palliative care recommendations are measured using Electronic Health Record [eHR] documentation of recommendations by hospitalist/clinician at Day 7. Each item in the ESAS is scored using: 0-10 (0= no pain; 10= worst possible pain), yielding a total score between 0 and 90.
Time Frame: Day 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 94 | 91
score on a scale | 28.7 (1.5) | 24.9 (1.5)

9. Other Pre Specified Outcome: Exploratory Aim 1b. Patient Symptom Burden (Edmonton Symptom Assessment Scale [ESAS])
Description: Patient symptom burden measured by Edmonton Symptom Assessment Scale [ESAS] mediated and/or moderated by patient/caregiver implementation of palliative care recommendations. Patient/caregiver implementation of palliative care recommendations are measured using patient/caregiver report at Day 7. Each item in the Edmonton Symptom Assessment Scale [ESAS] is scored using: 0-10 (0= no pain; 10= worst possible pain), yielding a total score between 0 and 90.
Time Frame: Day 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
score on a scale | 24.9 (1.5) | 28.7 (1.5)

10. Other Pre Specified Outcome: Exploratory Aim 1c. Caregiver Burden (Montgomery Borgatta Caregiver Burden Scale [MBCB]).
Description: Caregiver burden measured by Montgomery Borgatta Caregiver Burden Scale [MBCB] mediated and/or moderated by hospitalist/clinician implementation of palliative care recommendations. Implementation of palliative care recommendations are measured using Electronic Health Record [eHR] documentation of recommendations by hospitalist/clinician at Day 7. This scale contains a total of 14 questions and 5 Likert scale responses (a lot less, a little less, the same, a little more, or a lot more) with higher scores indicating greater burden. Caregiver burden will be quantified by three subscales; objective, subjective and demand burdens. Objective burden is measured by 6 questions (total score between 0-30), subjective burden is measured by 4 questions (total score between 4-20), and demand burden is measured by 4 questions (total score between 4-20).
Time Frame: Day 7
Population: Some participants did not answer which resulted in missing data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
score on a scale
  Objective Subscale: number analyzed (Participants) | 88 | 93
  Objective Subscale | 19.1 (0.3) | 19.4 (0.3)
  Subjective Subscale: number analyzed (Participants) | 78 | 85
  Subjective Subscale | 11.9 (0.3) | 11.6 (0.3)
  Demand Burden: number analyzed (Participants) | 72 | 78
  Demand Burden | 11 (0.3) | 10.8 (0.3)

11. Other Pre Specified Outcome: Exploratory Aim 1d. Caregiver Burden (Montgomery Borgatta Caregiver Burden Scale [MBCB]).
Description: Caregiver burden measured by Montgomery Borgatta Caregiver Burden Scale [MBCB] mediated and/or moderated by caregiver/patient implementation of palliative care recommendations. Caregiver/patient implementation of palliative care recommendations are measured using caregiver/patient report at Day 7. This scale contains a total of 14 questions and 5 Likert scale responses (a lot less, a little less, the same, a little more, or a lot more). Caregiver burden will be quantified by three subscales; objective, subjective and demand burdens. Objective burden is measured by 6 questions (total score between 0-30), subjective burden is measured by 4 questions (total score between 4-20), and demand burden is measured by 4 questions (total score between 4-20). Higher scores indicates greater burden.
Time Frame: Day 30
Population: Some participants did not answer which resulted in missing data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 105 | 104
score on a scale
  Objective burden: number analyzed (Participants) | 86 | 91
  Objective burden | 19.4 (0.3) | 19.1 (0.3)
  Subjective Burden: number analyzed (Participants) | 72 | 87
  Subjective Burden | 11.8 (0.3) | 12.2 (0.3)
  Demand Burden: number analyzed (Participants) | 68 | 79
  Demand Burden | 11.3 (0.3) | 11.3 (0.3)

12. Other Pre Specified Outcome: Exploratory Aim 1e. Caregiver Evaluation of Quality of End-of-Life Care [CEQUEL]
Description: Caregiver evaluation of end-of-life care quality measured by Caregiver Evaluation of Quality of End-of-Life Care [CEQUEL]
Time Frame: 2-3 Months after death of patient, if applicable
Population: This data was not collected.
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Exploratory Aim 1f. Caregiver Bereavement (Caregiver Bereavement Items ([CBI])
Description: Caregiver bereavement measured by Caregiver Bereavement Items ([CBI]
Time Frame: 2-3 Months after death of patient, if applicable
Population: This was not collected.
Arm/Group | Active Intervention | Usual Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Only patients were in both active intervention and usual care were monitored for adverse events. Caregivers were not monitored.
Groups:
- Active Intervention/Patients Only: Usual Care + Tele-consult Intervention
  Active Intervention: Half of the patients will receive tele-consult program. Tele-consult intervention includes: initial consult and 2 follow up contacts. Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
- Usual Care/Patients Only: Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
  Usual Care: Half of the patients will receive usual care. Usual care includes assessment and treatment by the admitting physician, along with any subspecialists that are consulted.
Arm/Group | Active Intervention/Patients Only | Usual Care/Patients Only
All-Cause Mortality (participants affected / at risk) | 2/105 | 2/104
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/104
Other Adverse Events (participants affected / at risk) | 0/105 | 0/104

LIMITATIONS AND CAVEATS:
The hospital sites restricted recruitment practices due to COVID-19. Therefore, recruitment was delayed one year. The delay resulted in not reaching the target number of participants. We reached saturation at 209 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT03767517/Prot_SAP_000.pdf